CLINICAL TRIAL: NCT02252198
Title: Evaluation of Non-Inferiority of Two Fast Follower Nucleic Acid Amplification Tests for the Diagnosis of Pulmonary Tuberculosis in Comparison to Geneexpert MTB/RIF
Brief Title: Evaluation of Non-Inferiority of Two Fast Follower Nucleic Acid Amplification Tests
Acronym: FIND
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Boston Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00085221; NA_00085221 (Other: Johns Hopkins University)
Record Dates: First submitted 2014-09-23; First posted 2014-09-30 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Investigational: • Participants will be asked to provide a total of three sputum samples over Days 1 and 2. The intent is for all samples to be collected before the subject starts any form of TB treatment. The first specimen (S1) should be 2 ml or greater in volume, and the second and third specimens (S2 and S3) should each be 1 ml or greater in volume. On Day 1, each participant will be asked to submit one spot sputum (S1) after enrollment and a second spot sputum after at least 2 hours (S2). Participants will be instructed to come back the following day (Day 2) and provide a third spot sputum (S3). In the event that a participant fails to return on Day 2, S3 may be collected a maximum of 7 days after enrollment, provided that no TB treatment has been initiated.
  Interventions: Other: Epistem Genedrive® and MolBio Truenat™

INTERVENTIONS:
Other: Epistem Genedrive® and MolBio Truenat™ — S1 will undergo direct smear and Epistem Genedrive® (optional for phase 2*) testing, before being homogenized with glass beads and split into three portions for testing with Epistem Genedrive®, MolBio Truenat™ and GeneXpert MTB/Rif® respectively. S2 and S3 will be randomized as to the order of testing using Epistem Genedrive® and MolBio Truenat™.

SUMMARY:
Assess sensitivity and specificity of two nucleic acid amplification tests, namely Epistem Genedrive® and MolbioTruenat™ in raw sputum compared to the WHO-endorsed GeneXpert® MTB/RIF assay using a gold standard of four cultures

DETAILED DESCRIPTION:
* Estimate the accuracy of the Epistem Genedrive® and MolbioTruenat™ in raw sputum and in sputum pellets.
* Assess the operational feasibility of Epistem Genedrive® and MolbioTruenat™
* Determine and compare costs between the Epistem Genedrive®, MolbioTruenat™, and Xpert MTB/RIF tests

ELIGIBILITY:
Inclusion Criteria:

* • Clinical suspicion of pulmonary TB (including cough ≥2 weeks and at least 1 other symptom typical of TB);

  * Age 18 years or above;
  * Willingness to have a study follow-up visit, if necessary, approximately two months after enrollment
  * Willingness to provide 3 sputum specimens at enrollment
  * Provision of informed consent.

Exclusion Criteria:

* • Receipt of ≥48 cumulative hours OR three or more doses of anti-TB treatment (defined as combination anti-TB therapy intended to treat active TB) within 60 days prior to completion of sputum collection;

  * Inability to provide informed consent (e.g. mentally impaired)
  * Enrolled individuals who do not provide a first sputum sample of ≥ 2ml and a second and third sputum sample of ≥ 1ml each will be classified as early exclusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with clinical suspicion of pulmonary TB.
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of tests | 4 months
  Non-inferiority of Epistem Genedrive® MTB iD Test and MolBio Truenat™ TB Assay to GeneXpert MTB/RIF using a non-inferiority margin of 5% for sensitivity in smear-positive, culture-positive; 7% for overall C+ sensitivity; and 3% for specificity in smear-negative, culture-negatives
Sensitivity and specificity of Epistem Genedrive® MTB iD | 4 months
  Sensitivity and specificity of Epistem Genedrive® MTB iD Test on raw sputum before homogenization, homogenized raw sputum and sputum pellet against a gold standard of concentrated smear and four cultures.
Sensitivity and specificity of MolBio Truenat™ TB Assay | 4 months
  Sensitivity and specificity of MolBio Truenat™ TB Assay on homogenized raw sputum and sputum pellet against a gold standard of concentrated smear and four cultures.

SECONDARY OUTCOMES:
Failure rate for the Epistem Genedrive® system assay and for the MolBio Truenat™ assay | 10 months
  Failure rate for the Epistem Genedrive® system assay and for the MolBio Truenat™ assay, expressed as the proportion of tests that require repeating due to an indeterminate or uninterpretable initial result (separately and together for tests performed on raw sputum and sputum pellet
Training needs for each assay | 10 months
  Training needs for each assay assessed objectively by number of hours of training, number of runs required, and successful completion of a proficiency assessment by trainees; training needs also will be assessed subjectively by the trainers and by user questionnaires
Operational feasibility | 10 months
  Operational feasibility will be assessed according to the infrastructure required to support each test, the robustness of the reagents and equipment (any breakdowns, storage requirements or contamination events), and the time it takes to run each test;
Cost-comparison between assays | 10 months
  A cost-comparison between assays assessing the cost per sample run incorporating all costs involved in transport, equipment, reagents, personnel, etc. will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Inbaraj LR, Daniel J, Sathya Narayanan MK, Srinivasalu VA, Bhaskar A, Scandrett K, Rajendran P, Kirubakaran R, Shewade HD, Malaisamy M, Padmapriyadarsini C, Takwoingi Y. Truenat MTB assays for pulmonary tuberculosis and rifampicin resistance in adults and adolescents. Cochrane Database Syst Rev. 2025 Mar 24;3(3):CD015543. doi: 10.1002/14651858.CD015543.pub2. PMID 40122135